CLINICAL TRIAL: NCT05509361
Title: An Open-label, Single-arm, Multi-center Study to Evaluate the Long-term Safety and Efficacy of AK101 Injection in Subjects With Moderate-to-severe Plaque Psoriasis
Brief Title: Open Label Study to Evaluate the Safety and Efficacy of AK101 Injection Subcutaneously in Subjects With Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK101-303
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK101 135mg (Experimental): Subjects who have completed AK101-302 receive AK101 135mg injection subcutaneously every 12 weeks.
  Subjects newly enrolled receive AK101 135mg injection subcutaneously at Week 0, 4 and then every 12 weeks.
  Interventions: Biological: AK101 injection SC

INTERVENTIONS:
Biological: AK101 injection SC — AK101 is supplied as 135 mg doses, provided in 1 mL prefilled syringes.

SUMMARY:
This is an open-label Phase III clinical study to evaluate the long-term safety and efficacy of AK101 injection in subjects with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
This is an open-label, single-arm, multi-center phase III study. The purpose of this study is to evaluate the long-term safety and efficacy of AK101 injection in subjects with moderate-to-severe plaque psoriasis. Subjects who have completed the previous Akeso registration trial with AK101 injection (AK101-302) and subjects who are to be newly enrolled will both receive AK101 135mg injection subcutaneously.

ELIGIBILITY:
Key Inclusion Criteria:

* Applicable for subjects who have completed the previous Akeso trial (AK101-302) with AK101 injection:

  1. Subjects can continue to participate in this study based on assessment of investigator.
  2. Subjects voluntarily participate in this study.
  3. Subjects who are women of childbearing potential must be practicing an adequate, medically acceptable method of birth control during the treatment period and for at least 6 months after the last study drug administration.
* Applicable for subjects newly enrolled:

  1. Male or female subjects aged ≥ 18 years old.
  2. Subjects diagnosed with moderate-to-severe plaque psoriasis and are applicable to systematic treatment.
  3. At screening and baseline, PASI score ≥ 12, Body Surface Area BSA (BSA) ≥ 10%, sPGA ≥ 3.
  4. Subjects who are applicable for biological agents, based on the assessment of investigator.
  5. Subjects who are women of childbearing potential must have a negative pregnancy test at screening and must be practicing an adequate, medically acceptable method of birth control for at least 6 months after the last study drug administration.

Key Exclusion Criteria:

* Applicable for subjects who have completed the previous Akeso trial (AK101-302) with AK101 injection:

  1. Subjects who have severe AE or SAE occurred in an Akeso trial with AK101 injection.
  2. Subjects who used prohibited drugs in an Akeso trial with AK101 injection.
  3. Subjects performed poor compliance in an Akeso trial with AK101 injection, based on the assessment of investigator.
  4. Subjects with any other disease, abnormal physical examination or abnormal laboratory examination leading to inapplicable for participating this study, based on the assessment of investigator.
* Applicable for subjects newly enrolled:

  1. Forms of psoriasis other than chronic plaque-type psoriasis.
  2. History or evidence of active TB. Patients with evidence of latent tuberculosis may enter the trial after sufficient treatment had initiated and maintained according to protocol.
  3. Positive results of confirmatory test for hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or syphilis.
  4. History of repeated chronic infection, had any serious infection or systemic infection within 2 months before screening.
  5. History of prohibited psoriasis treatments within 2/4 weeks before randomization.
  6. History of IL-12/23 or IL-23 inhibitors therapy.
  7. Inadequate washout period of prior biological therapy.
  8. History of malignant tumour within 5 years before screening.
  9. Any medical or psychiatric condition, laboratory, or ECG parameter which, in the opinion of the Investigator would place the subject at risk, interfere with participation or interpretation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Occurrence of Treatment-Emergent Adverse Event | up to 52 weeks
  To evaluate long-term safety as assessed by occurrence of TEAE.

SECONDARY OUTCOMES:
Occurrence of Serious Adverse Event and Adverse Events of Special Interest | up to 52 weeks
  To evaluate long-term safety as assessed by occurrence of SAE and AESI.
Percentage of Subjects Who Achieved at least 50% (PASI 50), 75% (PASI 75) and 90% (PASI 90) Reduction in Psoriasis Area and Severity Index (PASI) Score | up to 52 weeks
  PASI is a combined assessment of a lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for a final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4).
  PASI 50, PASI75 and PASI 90 were defined as participants achieving >= 50%, >= 75% or >= 90% improvement from baseline, respectively.
Percentage of Subjects Who Achieved Static Physician Global Assessment (sPGA) Clear(0) or Almost Clear(1) | up to 52 weeks
  The sPGA is an instrument providing a subjective evaluation of the overall severity of psoriasis, based on severity of induration, scaling, and erythema. The scores are: 0 = clear; 1 = minimal; 2 = mild; 3 = moderate; 4 = marked; 5 = severe.
Pharmacokinetics Assessment of AK101 Serum Concentration | up to 52 weeks
Immunogenicity Assessment with Number and Percentage of Subjects with Detectable Anti-AK101 Antibody (ADA) | up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university people's hospital, Beijing, China